CLINICAL TRIAL: NCT01825174
Title: Musculoskeletal Consequences of Pediatric Overweight - Efficiency of Different Interventions on Health, Motor and Psychosocial Development in Overweight and Obese Children
Brief Title: Overweight Children - Musculoskeletal Consequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. med. Benita Kuni, MD, Orthopedic and Trauma Surgeon, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213-2006-130321
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Non-overweight children in ball games program (Active Comparator): twice a week different ball games 90min
  Interventions: Behavioral: Ball games program
- Overweight children in nutrition counseling program (Experimental): 9 units of 90min each of nutrition counseling
  Interventions: Behavioral: Nutrition counseling
- Control group overweight children (Placebo Comparator): No intervention during six months
- Overweight children in ball games program (Experimental): twice a week different ball games 90min
  Interventions: Behavioral: Ball games program
- Overweight children in ball games and nutrition counseling (Experimental): twice a week different ball games 90min and 9 units of 90min each of nutrition counseling
  Interventions: Behavioral: Ball games program; Behavioral: Nutrition counseling
- Non-overweight control (no intervention) (Placebo Comparator)

INTERVENTIONS:
Behavioral: Ball games program — twice a week different ball games 90min
  Arms: Non-overweight children in ball games program; Overweight children in ball games and nutrition counseling; Overweight children in ball games program
Behavioral: Nutrition counseling — 9 units of 90min each of nutrition counseling
  Arms: Overweight children in ball games and nutrition counseling; Overweight children in nutrition counseling program

SUMMARY:
The purpose was to investigate the consequences of pediatric overweight on the musculoskeletal system, postural control and proprioception, and to analyze prospectively the influence of ball games and nutrition counseling.

ELIGIBILITY:
Inclusion Criteria:

Overweight Children:

* BMI = or > than the gender, race, and age specific 92nd percentile from the National Children Health and Nutrition Examination Survey

All participants:

- 6-11 y. old

Exclusion Criteria:

* severe impairment with functional restriction of the upper or lower extremities (due to injuries)
* neurological deficits/diseases compromising the postural control
* important communication problems due to another mother language

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in error points in one legged-standing test | at baseline and 6 months later after intervention

SECONDARY OUTCOMES:
Change in angle deviation from target angle in angle reproduction test | at baseline and 6 months later after intervention
Change in range of motion at the joints of the lower extremities | at baseline and 6 months later after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schmitt, M.D. Ph.D., Principal Investigator — University of Heidelberg/ ATOS Clinic Heidelberg
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Kuni B, Ruhling NE, Hegar U, Roth C, Schmitt H. Ball games and nutrition counseling improve postural control in overweight children. BMC Pediatr. 2015 Dec 11;15:205. doi: 10.1186/s12887-015-0523-4. PMID 26654525